CLINICAL TRIAL: NCT07312266
Title: Questioning the Epidemiology of Asymptomatic TB
Acronym: TB QUEST
Status: Recruiting | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Responsible Party: Principal Investigator, Alberto Garcia-Basteiro, Research Professor, Barcelona Institute for Global Health
Other Study IDs: 101117940; ERC-2023-STG-101117940 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis; Tuberculosis (TB); HIV; HIV (Human Immunodeficiency Virus)
Keywords: Asymptomatic tuberculosis; Asymptomatic; Subclinical tuberculosis; Subclinical
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Sputum, tongue swabs, urine, stool, blood, saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic: Contacts of bacteriologically-confirmed asymptomatic TB index cases
- Symptomatic: Contacts of bacteriologically-confirmed symptomatic TB index cases

SUMMARY:
Tuberculosis (TB) remains one of the world's leading causes of morbidity and mortality. Current TB control strategies focus largely on the binary paradigm of TB, which tackle Mtb infection and the symptomatic stages of the disease as the major drivers of the TB epidemic. However, prevalence surveys have shown that about 50% of cases in which Mycobacterium tuberculosis is isolated from sputum but do not report having symptoms. Therefore, asymptomatic TB may play an important role in TB transmission. However, no field study has demonstrated direct transmission from a subclinical TB case to a confirmed secondary case.

TB-QUEST is an ERC-funded epidemiological field study that aims to provide direct evidence of effective transmission from asymptomatic TB cases to their close contacts using advanced genomic methods, and to better characterize the asymptomatic stage of TB within the natural history of disease.

DETAILED DESCRIPTION:
The majority of TB control policies rely on the binary paradigm of 'latent' and 'active' TB. Recent research demonstrates that TB exists on a continuous spectrum of bacterial and immunological responses, and sheds light on the non-linear path that TB may take to advance or regress along the spectrum of disease. This understanding has led to the distinction between latent (M.tb infection), asymptomatic, and active (symptomatic) TB stages. Asymptomatic TB (aTB) stages have attracted increased scientific interest since they could play an important role in TB transmission. If this were the case, the implications for global TB control and research would be enormous. Thus, there is an urgent need for intensified research into this TB stage to better understand its public health importance and implications on TB transmission.

TB QUEST is a prospective epidemiological field study designed to address several critical research gaps surrounding aTB. The overall aim of the study is to provide direct evidence of asymptomatic TB transmission, and to better characterize the asymptomatic TB stage within the natural history of disease. This project has four main objectives:

Objective 1: To provide direct evidence on the successful transmission of tuberculosis infection (leading to TB disease) by individuals diagnosed with aTB Objective 2: To ascertain the presence of typical TB symptoms in self-reported asymptomatic laboratory-confirmed TB patients Objective 3: To understand the factors associated with Mtb self-clearance or disease progression in patients with aTB Objective 4: To understand the characteristics and progression of non-infectious aTB

TB QUEST will recruit asymptomatic and symptomatic index TB cases as well as their close contacts, allowing for the observation of secondary (genomically-linked) cases and new infections while providing direct temporal characterization and directionality of TB transmission. In addition, TB QUEST nests three additional longitudinal assessments among individuals with aTB in order to ascertain presence of symptoms and assess their clinical trajectory.

The project is coordinated by the Barcelona Institute for Global Health (ISGlobal) in close collaboration with the Centro de Investigação em Saúde de Manhiça (CISM), located in the district of Manhiça, Mozambique, where all field work will be conducted. The district of Manhiça is a high TB/HIV burden area in Southern Mozambique, where the latest reported TB case notification is around 500 per 100,000 population and the prevalence of HIV in the adult population was 35%.

TB QUEST will conduct an initial cross-sectional assessment among PLHIV attending routine follow up visits in order to identify bacteriologically-confirmed asymptomatic and symptomatic TB cases. It follows with a nested prospective contact cohort study in which two cohorts of close-contacts exposed to the aTB and clinical TB cases, respectively, will be followed up periodically for 12 months. The project embeds three additional longitudinal assessments: a) one among both asymptomatic and symptomatic TB cases to objectively verify the presence of common TB symptoms, b) one among a proportion of aTB cases that will be closely monitored for radiological, microbiological and clinical changes to assess the trajectory of aTB, and c) one in which a subset of non-infectious aTB patients will be followed to observe its trajectory.

TB-QUEST will generate high-quality evidence to resolve the current hypotheses on aTB transmission. If aTB plays and important role in TB transmission, the current pillars of TB control will prove to be insufficient to achieve the reduction of TB incidence and mortality set by the international community. Thus, this proposal has the potential to represent a paradigm shift for TB control. The evidence derived from this study will challenge global symptom-driven case finding strategies, as well as the clinical management of aTB cases. Further, disentangling the evolution of aTB may allow for its inclusion as a primary endpoint in TB vaccine and drug trials, improving efficiency in future TB research and the development of new tools to fight the disease.

ELIGIBILITY:
Index cases:

Inclusion Criteria:

1. 18 years of age or older
2. Documented HIV infection
3. Presenting at a health facility for routine HIV care

Exclusion Criteria:

1. History of TB treatment in the last 12 months
2. Pregnant women
3. Refusal to provide consent for study procedures
4. Contra-indication to any sampling procedure required by the study

Study 3 will utilize additional inclusion criteria:

Inclusion criteria:

1. On ART for less than 6 months
2. No evidence of viral suppression
3. Documented CD4 count >350 copies/ul
4. TB-suggestive x-ray
5. Verified absence of fever and cough, as ascertained through the symptom trackers

Contacts:

Inclusion criteria: All close contacts (household and close community contacts) will be offered to participate in the study, regardless of age or HIV status.

Exclusion criteria:

1. Plans to migrate in the next 12 months
2. Pregnant women
3. Currently taking anti-tuberculosis treatment or preventive TB treatment
4. Contacts with co-prevalent TB identified at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants attending routine HIV care at the Manhica District Hospital
Sampling Method: Non-Probability Sample
Enrollment: 6770 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of secondary cases arising from TB index case transmission | 12 months
  Transmission from aTB cases will be compared to that of clinical cases by: i) comparing the proportion of genomically-linked secondary cases and ii) by comparing the proportion of QFT conversion and host transcriptomic changes

SECONDARY OUTCOMES:
Symptomatology of asymptomatic TB | 2 weeks
  The objectively measured frequency of symptoms among asymptomatic TB cases compared to that of symptomatic TB cases
Clinical trajectory of aTB | 12 months
  The proportion of aTB cases with measurable signs of progression to symptomatic or worsening TB disease compared to those who self-clear.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigação em Saúde de Manhiça (CISM), Manhiça, Maputo Province, Mozambique

IPD SHARING:
Plan to Share IPD: Undecided